CLINICAL TRIAL: NCT04533490
Title: A Multi-center, Single-arm, Open Phase Ⅱ Clinical Trial of Camrelizumab for Adjuvant Treatment of Resectable Esophageal Squamous Cell Carcinoma
Brief Title: A Phase Ⅱ Clinical Trial of Camrelizumab for Adjuvant Treatment of Resectable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, DOCTOR, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-123
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Resectable Esophageal Squamous Cell Carcinoma
Keywords: ESCC,Adjuvant therapy,Camrelizumab
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 (Experimental): After the subjects were enrolled in the study, the patients were treated with SHR-1210 (200mg ivgtt q3w) from 1 to 2 months after operation until disease progression or intolerable toxicity, and the longest medication period was no more than 12 months
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — After the subjects were enrolled in the study, the patients were treated with SHR-1210 200mg igvtt q3w from 1 to 2 months after operation until disease progression or intolerable toxicity, and the longest medication period was no more than 12 months

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of SHR-1210 for adjuvant treatment of resectable esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
Although esophagectomy is still the standard treatment for patients with localized esophageal cancer, the long-term therapeutic effect is not satisfactory.About 50% of patients experienced relapse in the first year after treatment. The 5-year survival rate of esophageal cancer patients treated by surgery is still less than 30%. Although the effect of preoperative treatment is relatively clear, the effect of postoperative treatment, especially postoperative chemotherapy, is still controversial and no consensus has been reached.The basic reason is that the postoperative trauma of esophageal cancer is large, and the patients' tolerance to chemotherapy is poor. The efficacy of immunocheckpoint inhibitors in metastatic ESCC has been recognized.We plan to conduct a phase II multicenter, single arm, open phase II clinical trial to evaluate the efficacy and safety of humanized anti PD-1 monoclonal antibody SHR-1210 in adjuvant treatment of resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histology confirmed as esophageal squamous cell carcinoma;
2. The clinical stages are cT1b-T4aN0M0, cT1-T4aN+M0;
3. The subjects were required to complete preoperative concurrent chemoradiotherapy and complete R0 resection before enrollment;
4. The shortest time of neoadjuvant therapy was 6 weeks and the longest was 12 weeks;
5. Postoperative pathology: T1 or above T1, N1 or N1 above, no distant metastasis;
6. Aged 18-75;
7. ECOG:0-1;
8. The main organs function normally, that is, the following criteria are met:

   Blood routine examination:

   HB≥90g/L; ANC ≥ 1.5 × 109 / L; PLT ≥ 80 × 109 / L;

   Biochemical examination:

   ALB ≥ 30g / L;b.ALT and AST ≤ 2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN;c.TBIL ≤ 1.5ULN;d.plasma Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min;
9. There was no serious concomitant disease with a survival time of less than 5 years;
10. Voluntary and able to comply with the protocol during the study;
11. Provide written informed consent before entering the study, and patients have understood that they can withdraw from the study at any time without any loss.

Exclusion Criteria:

1. Patients with previous or concurrent malignant tumors, except for skin basal cell carcinoma and cervical carcinoma in situ that have been cured; patients with small gastric stromal tumor and other tumors, which are judged by researchers to have no impact on the patient's life in the short term, can be excluded;
2. Participated in other drug clinical trials within four weeks;
3. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis,Hyperthyroidism; patients with vitiligo ; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
4. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppressive purposes (dose> 10 mg/day of prednisone or other therapeutic hormones) and continues to be used for 2 weeks prior to enrollment;
5. Any active malignant tumor within 2 years, except for the specific cancer under study in this study and locally recurrent cancer that has been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast cancer in situ);
6. Patients with known history of CNS metastasis or CNS metastasis before screening. For patients with clinically suspected CNS metastasis, CT or MRI must be performed within 28 days before randomization to exclude CNS metastasis;
7. Patients with unstable angina pectoris history, newly diagnosed angina pectoris within 3 months before screening or myocardial infarction events occurred within 6 months before screening; arrhythmias (including QTCF: male ≥ 450 ms, female ≥ 470 MS) need long-term use of antiarrhythmic drugs and NYHA grade ≥ II cardiac insufficiency;
8. Urine routine examination showed that urinary protein was ≥ + +, and 24-hour urinary protein was more than 1.0 G;
9. For female subjects: they should be surgical sterilization, postmenopausal patients, or agree to use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period; the serum or urine pregnancy test must be negative within 7 days before the study enrollment, and must be non lactation period. Male subjects: they should be surgical sterilization or agree to use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period;
10. The patient had received liver transplantation;
11. Patients with infectious pneumonia, non infectious pneumonia, interstitial pneumonia and other patients who need to use corticosteroids;
12. Have a history of chronic autoimmune diseases, such as systemic lupus erythematosus, etc;
13. Patients had a history of inflammatory bowel disease such as ulcerative enteritis and Crohn's disease, and a history of chronic diarrhea such as irritable bowel syndrome;
14. Patients with a history of sarcoidosis or tuberculosis;
15. Patients with a history of active hepatitis B and hepatitis C and HIV infected patients;
16. Patients with a history of psychotropic substance abuse and can't quit or have mental disorders;
17. Pleural effusion or ascites with clinical symptoms and requiring clinical intervention;
18. Patients with a history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
19. According to the judgment of the researchers, there are accompanying diseases that seriously endanger the safety of patients or affect patients to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
RFS(relapse free survival) | up to 1 year
  Recurrence free survival of resectable esophageal squamous cell carcinoma treated with SHR-1210
DFS（disease-free survival） | up to 1 year
  Disease-free survival of resectable esophageal squamous cell carcinoma treated with SHR-1210

SECONDARY OUTCOMES:
OS（overall survival rate） | At time of surgery
  From date of randomization until the date of death from any cause; Overall survival rate of resectable esophageal squamous cell carcinoma treated with SHR-1210

OTHER OUTCOMES:
Exploratory analysis of biomarkers for predicting efficacy | At time of surgery
  The relationship between PD-L1 dynamic expression, ctDNA sequencing and therapeutic effect was evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University